CLINICAL TRIAL: NCT00005265
Title: Natural History of Coronary Heart Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1149; R03HL045495 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2001-11

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Myocardial Infarction; Heart Diseases; Death, Sudden, Cardiac; Heart Failure, Congestive; Heart Failure
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Myocardial Infarction; Heart Diseases; Death, Sudden, Cardiac; Heart Failure

SUMMARY:
To examine the natural history of mortality due to coronary heart disease in post-myocardial infarction patients from the Beta-Blocker Heart Attack Trial (BHAT) and the Aspirin Myocardial Infarction Study (AMIS).

DETAILED DESCRIPTION:
BACKGROUND:

In January 1990, the National Heart, Lung, and Blood Institute issued a Program Announcement establishing a Small Grants Program to provide limited support to extend analyses of research data generated by clinical trials, population research, and demonstration and education studies. This study used data collected in two completed clinical trials, the BHAT and AMIS.

DESIGN NARRATIVE:

Study endpoints included all-cause mortality, cause-specific mortality such as sudden death, recurrent and non-fatal myocardial infarction, and incident congestive heart failure. Univariate and multivariate analyses of baseline data variables from BHAT were conducted to determine which were predictive of study endpoints. Baseline variables included sociodemograhic characteristics, medical history, medication use, physical examination finds, and electrocardiographic characteristics. Baseline characteristics found to be predictive of study endpoints in the BHAT placebo group were examined in the AMIS placebo group. Long- and short-term prognoses for patients suffering a transmural myocardial infarction were compared for those suffering a subendocardial infarction.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1990-09; Study Completion 1992-05 (Actual)